CLINICAL TRIAL: NCT06121674
Title: Shaeer's Vein Ligation - II: Internal Pudendal Vein Perineal Ligation For The Management of Veno Occlusive Erectile Dysfunction. The Surgical Study
Brief Title: Shaeer's Vein Ligation-II: Internal Pudendal Vein Perineal Ligation For Veno Occlusive Erectile Dysfunction
Acronym: Shaeer-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Osama Shaeer, Prof.Dr.Osama Shaeer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shaeer's Vein Ligation-II
Record Dates: First submitted 2023-11-01; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Erectile Dysfunction; Erectile Dysfunction Due to Venous Disorder
Keywords: veno-occlusive erectile dysfunction; erectile dysfunction; venous leak; internal pudendal vein ligation
MeSH Terms: conditions — Erectile Dysfunction | interventions — Penile Implantation

STUDY DESIGN:
Intervention Model Description: Surgery shall be performed for patients with VOD who are not responding to medical treatment and are candidate for penile prosthesis implantation. VOD will be documented by cavernosography to affect the deep system of veins; the internal pudendal vein, unilaterally.
  Patients will be randomized into two groups: one to proceed to Penile Prosthesis Implantation (PPI Group), and another to be offered a choice between PPI or SHAEER-II. Patients opting for PPI will be assigned to the PPI group. Patients opting to SHAEER-II will be assigned to (SHAEER-II group).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shaeer-II (Experimental): SHAEER-II targets ligation of the internal pudendal vein at the point where the vein exits Alcock's canal, and courses lateral to the ischial tuberosity.
  Patient is oriented in the lithotomy position. The ischial tuberosity is marked. An incision is cut medial to the ischial tuberosity. Subcutaneous fat is dissected down to the neurovascular bundle harboring the internal pudendal vein. The vein is then ligated.
  Interventions: Procedure: Shaeer-II
- PPI (Active Comparator): Penile prosthesis implantation (PPI) will be performed
  Interventions: Procedure: PPI

INTERVENTIONS:
Procedure: Shaeer-II — SHAEER-I targets ligation of the internal pudendal vein at the point where the vein exits Alcock's canal, and courses lateral to the ischial tuberosity.
  Patient is oriented in the lithotomy position. The ischial tuberosity is marked. An incision is cut medial to the ischial tuberosity. Subcutaneous fat is dissected down to the neurovascular bundle harboring the internal pudendal vein. The vein is then ligated.
  Other Names: Shaeer's Vein Ligation - II; Internal Pudendal Vein Perineal Ligation
  Arms: Shaeer-II
Procedure: PPI — Penile Prosthesis Implantation will be performed
  Other Names: Penile Prosthesis Implantation
  Arms: PPI

SUMMARY:
The goal of this interventional study is to evaluate a new surgical technique (Shaeer's Perineal Internal Pudendal Vein Ligation (SHAEER-II)) in patients with deep system veno-occlusive erectile dysfunction (VOD)

. The main question[s] it aims to answer are:

* [Will the patients have satisfactory rigidity after surgery]
* [What will the Satisfaction rates be]
* [Will there be complications]

Participants will

* Undergo SHAEER-II or PPI surgery
* Report the results of surgery for at least 6 months

DETAILED DESCRIPTION:
Title Shaeer's Vein Ligation - II: Internal Pudendal Vein Perineal Ligation For The Management of Veno Occlusive Erectile Dysfunction. The Surgical Study

Objectives Vein ligation surgery for veno-occlusive erectile dysfunction (VOD) has largely been unsuccessful, possibly due to the extensive collateral circulation, but also due to confinement to intermediate vein system ligation. The deep system of veins has been surgically inaccessible.

This is study evaluates Shaeer's Vein Ligation - II (Shaeer-II): a surgical technique for ligation of the deep system of veins; the internal pudendal vein.

Methods Surgery shall be performed for patients with VOD who are not responding to medical treatment and are candidate for penile prosthesis implantation. VOD will be documented by cavernosography to affect the deep system of veins; the internal pudendal vein, unilaterally.

Patients will be randomized into two groups: one to proceed to Penile Prosthesis Implantation (PPI Group), and another to be offered a choice between PPI or SHAEER-II. Patients opting for PPI will be assigned to the PPI group. Patients opting to SHAEER-I will be assigned to (SHAEER-II group).

Primary outcome will be measured as per satisfaction rates and erectile function, at the 6th month post-operative. Evaluation shall be through the Treatment Satisfaction Scale (TSS) Scores and the Abbreviated International Index of Erectile Function (IIEF-5). Outcome assessor/s shall be blinded as to the patient group. Secondary outcome will be complications -if any.

Surgical Technique for SHAEER-II:

SHAEER-II targets ligation of the internal pudendal vein at the point where the vein exits Alcock's canal, and courses lateral to the ischial tuberosity.

Patient is oriented in the lithotomy position. The ischial tuberosity is marked. An incision is cut medial to the ischial tuberosity. Subcutaneous fat is dissected down to the neurovascular bundle harboring the internal pudendal vein. The vein is then ligated.

Pre-operative Evaluation:

* Patients will fill the IIEF-5 questionnaire
* Review of past-utilization of medical treatment for ED (erectile dysfunction)
* Laboratory Investigations: serum testosterone (free and total), prolactin, blood sugar profile, lipid profile, general pre-operative investigations.
* Imaging: penile duplex and cavernosography.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with deep system veno-occlusive erectile dysfunction
* Lack of response to medical treatment for erectile dysfunction including PDEi (Phosphodiesterase Inhibitors), aphrodisiacs, hormonal therapy (if there is a hormonal disturbance), and intracavernous injections, despite control of risk factors such as diabetes mellitus.

Exclusion Criteria:

* Patients with uncontrolled diabetes, smokers and patients with anesthesia risk
* Patients with arteriogenic erectile dysfunction, penile fibrosis, Peyronie's disease or psychiatric disorders.
* Patients with bilateral deep system VOD
* Patients who refuse to participate in the study

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction Scale | 6 months
  A questionnaire to assess satisfaction with the results of surgery
Abbreviated International Index of Erectile Function | 6 months
  A questionnaire to assess erectile function

SECONDARY OUTCOMES:
Complications | 6 months
  Complications - if any - shall be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Osama Shaeer, MD,PhD, Study Chair — kasr El Aini Faculty of Medicine, Cairo University, Egypt
Locations (1):
- Kasr El Aini Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No